CLINICAL TRIAL: NCT07168785
Title: [18F]-AraG PET Imaging for Enhanced Risk Stratification and Chemoradiotherapy Response Assessment in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: [18F]-AraG PET Imaging in LA HNSCC
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: CellSight Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Langer, Professor of Clinical Radiation Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTO-IUSCCC-0910
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC); Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: AraG PET/CT; Chemoradiotherapy; [18F]-AraG PET/CT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- [18F]-AraG PET/CT scan (Experimental): [18F]-AraG PET/CT scans to be performed according to the institution's standard of operation, which occurs on the first and sixteenth day of treatment.
  Interventions: Drug: [18F]-AraG radiotracer; Drug: Chemotherapy; Device: Radiotherapy

INTERVENTIONS:
Drug: [18F]-AraG radiotracer — [18F]-AraG radiotracer, which occurs on the first and sixteenth day of treatment.
Drug: Chemotherapy — Concurrent chemoradiotherapy (CRT) with weekly doses of cisplatin.
Device: Radiotherapy — Concurrent chemoradiotherapy (CRT) of 70Gy of radiation dose in 33 fractions.

SUMMARY:
This study will use [18F]-AraG PET/CT scans to monitor patients who have been diagnosed with locally advanced Head and Neck Squamous Cell carcinoma (LA-HNSCC), and are planning to undergo standard of care chemoradiotherapy for treatment.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is the seventh most common cancer globally. Definitive chemoradiotherapy (CRT) remains the standard of care (SOC) treatment for LA-HNSCC, yet some patients are unsuccessfully treated. The purpose of this study is to explore the feasibility and possible function of [18F]-AraG PET/CT (a diagnostic procedure that uses a radioactive tracer [A method that uses radioactive substances to make pictures of areas inside the body] to image tumors and assess response to treatment) scans performed before and during treatment to monitor response in patients undergoing chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria

1. Patients ≥18 years of age.
2. Ability to provide written informed consent and HIPAA authorization.
3. LA-HNSCC in the larynx, hypopharynx, or human papillomavirus (HPV) negative oropharynx and is planning to receive definitive CRT as the SOC treatment, which includes a total of 70 Gy of radiation dose in 33 fractions, delivered over 5 days a week for 7 weeks, as well as planned weekly cycles of cisplatin (CDDP).
4. Tumor stage III and IV (AJCC 8th edition).
5. Unresectable cases.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Willing and able to maintain the imaging protocol.
8. Patients planning to receive pre-CRT and post-CRT FDG PET/CT scans as part of the standard clinical practice.

Exclusion Criteria

1. Diagnosis of immunodeficiency or receiving systemic steroid therapy or any form of immunosuppressive therapy within 7 days prior to the PET/CT scan.
2. Pregnant or breastfeeding.
3. Patients that will receive definitive induction chemotherapy or surgery.
4. Patients who are unable to complete the radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
[18F]-AraG PET/CT uptake and infiltrating cytotoxic T-cell expression. | Week 1 and Week 16
  Examining the distribution of [18F]-AraG PET SUV metrics and counts of CD3+/CD8+/PD1- and CD3+/CD8+/PD1+ T-cells
Pre-treatment [18F]-AraG PET/CT uptake and clinical response. | Pre-treatment
  Correlation of pre-treatment [18F]-AraG PET/CT metrics (such as SUVmax, mean and uptake volume) and clinical response.
Changes between pre-treatment and mid-treatment [18F]-AraG PET/CT uptake and clinical response | Pre-treatment and Week 16
  Correlation between percentage changes in PET uptake values (max, mean, and peak) at pre- and mid-CRT and treatment response categories.

SECONDARY OUTCOMES:
Individual cytotoxic T-cell activities (CD3+, CD8+, PD1-, and PD1+) and pre-treatment [18F]-AraG PET/CT uptake | Pre-Treatment
  Correlation between individual cytotoxic T-cell activities (CD3+, CD8+, PD1-, and PD1+) and pre-treatment [18F]-AraG PET/CT uptake.
Tumor extent and standard uptake values between FDG PET and [18F]-AraG PET/CT imaging | treatment planning through post treatment ( up to 6 months)
  Identify accuracy in tumor extent and standard uptake values between FDG PET and [18F]-AraG PET/CT imaging.
[18F]-AraG PET/CT uptake over time and progressive-free survival | up to 6 months
  Association between the pattern of change in [18F]-AraG PET/CT uptake over time and progressive-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Langer, Principal Investigator — Indiana University Simon Comprehensive Cancer Center
Locations (1):
- Indiana University, Indianapolis, Indiana, United States